CLINICAL TRIAL: NCT03512730
Title: BENEFITS OF A NEW MECHANICAL DECONTAMINATION METHOD, TI-BRUSH, ON THE ADJUNCT TREATMENT OF REGENERATIVE THERAPY OF PERI-IMPLANTITIS LESIONS: 12-MONTH OUTCOMES OF A RANDOMIZED CONTROLLED CLINICAL TRIAL
Brief Title: A NEW MECHANICAL DECONTAMINATION METHOD IN PERI-IMPLANTITIS, TI-BRUSH, A RANDOMIZED CONTROLLED CLINICAL TRIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Beatriz de Tapia, Associate professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PERECL-201305
Record Dates: First submitted 2018-04-27; First posted 2018-05-01 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Peri-Implantitis
Keywords: regenera
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titanium brush, H2O2 3%, plastic curettes (Experimental)
  Interventions: Device: Titanium brush; Other: Classic decontamination
- H2O2 3%, plastic curettes (Active Comparator)
  Interventions: Other: Classic decontamination

INTERVENTIONS:
Device: Titanium brush — a titanium brush will be tested as mechanical decontamination in regenerative treatment of peri-implantitis
  Arms: Titanium brush, H2O2 3%, plastic curettes
Other: Classic decontamination — Classic decontamination will be performed by means of H2O2 3% and plastic curettes

SUMMARY:
Objective:

The objective of this study was to evaluate a new mechanical method (Ti-Brush, Straumann, AG, Basel, Switzerland) of implant surface decontamination.

Material and methods:

A randomized double-blinded controlled clinical trial with a 1-year follow-up it is being carried out. After a hygienic phase, defects were randomly assigned to a control (n=18) or to a test group (n=18). In control group, implant surface was decontaminated both mechanically and chemically with 3% H2O2 and plastic ultrasonic scalers, respectively, while in test group Ti-Brush was added. Infrabony defects in both groups were regenerated with BoneCeramic (Straumann, AG, Basel Switzerland) and collagen barrier membrane Cytoplast (Osteogenics, Lubbock, United States). Clinical and radiographic parameters were measured at baseline, 6, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy or treated periodontal patients
* A good level of oral hygiene (Plaque Index ≤ 25%) (O'Leary et al., 1972).
* Presence of at least one titanium implant exhibiting peri-implantitis (peri-implant bone loss > 30% and Implant PPD ≥ 6 mm with bleeding and/or pus suppuration on probing)
* Osseous defect had to be circumferential, or present at least two walls and 3mm depth.
* Presence of >1 mm of keratinized peri-implant mucosa
* Absence of systemic diseases that could influence the outcome of the therapy.

Exclusion Criteria:

* Pregnant or lactating women
* Esthetically compromised patients
* Patients who received systemic antibiotics in the past 3 months or treatment of peri-implantitis in the last 12 months.
* Smokers of more than 10 cigarettes a day

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Evaluate probing pocket depth changes by decontamination of the implant surface with ultrasonics, 3% H2O2, and Ti-Brush™ at 6 and 12 months. | 6 and 12 months

IPD SHARING:
Plan to Share IPD: Undecided
The results obtained are expected to be published in both national and international journals. In addition, the results will be disseminated national and international scientific events.

REFERENCES:
- [Derived] de Tapia B, Ribeiro-Amaral T, Mor C, Nart J, Valles C. Peri-implantitis reconstructive treatment implementing a titanium brush: 5-year extension results from a randomized clinical trial. J Periodontol. 2025 Nov;96(11):1213-1226. doi: 10.1002/JPER.24-0673. Epub 2025 Mar 28. PMID 40153369